CLINICAL TRIAL: NCT06725069
Title: Effects of Neuromuscular Electrical Stimulation Applied to Agonist or Antagonist Muscles of the Upper Extremity on Flexor Spasticity and Function in Patients With Stroke
Brief Title: Effects of Neuromuscular Electrical Stimulation on Flexor Spasticity and Function in Stroke Patients
Status: Completed | Type: Observational
Sponsor: Gaziler Physical Medicine and Rehabilitation Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Emrah Karaduman, Resident Doctor, Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Other Study IDs: E2-24-9437
Record Dates: First submitted 2024-12-01; First posted 2024-12-10 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-12

CONDITIONS: Stroke; Spastic Hemiplegia
Keywords: stroke; neuromuscular electrical stimulation; rehabilitation; hemiplegia; spasticity
MeSH Terms: conditions — Stroke; Hemiplegia; Muscle Spasticity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Agonist NMES: In the first group, NMES (Group 1=Agonist group) was applied to the wrist and finger flexors for 20 minutes in addition to conventional treatment.
  Interventions: Other: Neuromuscular Electrical Stimulation
- Antagonist NMES: In the second group, NMES (Group 2=Antagonist group) was applied to the wrist and finger extensors for 20 minutes in addition to conventional treatment.
  Interventions: Other: Neuromuscular Electrical Stimulation
- Exercise: Patients in the third group (Group 3=Control group) were included in an occupational rehabilitation program for 20 minutes to improve upper extremity functions in addition to conventional treatment.
  Interventions: Other: Control (Standard treatment)

INTERVENTIONS:
Other: Neuromuscular Electrical Stimulation — NMES was performed using the Enraf Nonius Myomed 632X device. Both applications were performed 5 days/week for 4 weeks. NMES was performed with the patients in a sitting position and the affected arm resting on a table with the forearm supinated (Agonist group) / forearm pronated (Antagonist group). Surface electrodes (50x50 mm self-adhesive) were placed on the wrist and finger flexor/extensor muscle group. NMES parameters; Symmetric biphasic, pulse width 200 μs, on time 6 seconds (ramp up 1 second, ramp down 2 seconds), off time 12 seconds, stimulation intensity according to the patient's tolerance (not exceeding 90 mA), frequency 50 Hz and was adjusted to elicit contraction in the flexor and extensor muscles of the wrist and fingers.
  Groups: Agonist NMES; Antagonist NMES
Other: Control (Standard treatment) — In addition to conventional treatment, participants were included in an occupational rehabilitation program for 20 minutes to improve upper extremity functions.
  Groups: Exercise

SUMMARY:
In this study, the investigators aimed to determine the effects of botulinum neurotoxin type A injections for wrist and finger flexor spasticity and neuromuscular electrical stimulation therapy applied to wrist and finger flexors or extensors on upper extremity flexor spasticity and function in stroke patients.

DETAILED DESCRIPTION:
Neuromuscular electrical stimulation therapy applied to wrist and finger flexors (agonist application) or wrist and finger extensors (antagonist application) after botulinum neurotoxin type A injections in stroke patients with wrist and finger flexor spasticity in upper extremity flexor spasticity, To determine the effects on motor recovery, upper extremity and hand functions, hand grip strength, range of motion, functional independence, quality of life, hand skills and sonographically evaluated muscle thickness and to compare these different applications.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with ischemic or hemorhagic stroke after imaging with CT/MRI
2. First time stroke survivor
3. between 45-75 years old
4. Stroke duration > 3 months
5. Neurologically stable
6. Affected wrist and finger flexor muscle spasticity with MAS≥2
7. Patients whose cognitive status is at a level to understand the study instructions MMT> 23)

Exclusion Criteria:

1. Presence of another neurological disorder other than stroke causing motor impairment/spasticity
2. Fixed contracture in the hand-wrist
3. Use of medical treatment for spasticity
4. Having received neurolytic therapy, BoNT-A injection or NMES treatment in the last 3 months
5. Skin problem (disease, allergy, infection, etc.) on the contact surface of the NMES
6. Complex regional pain syndrome (CRPS), sequelae of previous trauma or surgery (muscle tendon adhesion, peripheral nerve damage) in the affected extremity
7. Having a pacemaker
8. Epilepsy
9. Malignancy

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed with ischemic or hemorhagic stroke after imaging with CT/MRI
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2025-01-14 (Actual)

PRIMARY OUTCOMES:
The Modified Ashworth Scale (MAS) | Assessments will be conducted immediately before the treatment starts and at the end of the treatment (week 4).
  The Modified Ashworth Scale (MAS) is a clinical tool used to assess spasticity, which is characterized by increased muscle tone and resistance to passive movement. It is commonly applied in individuals with neurological conditions such as stroke, multiple sclerosis, or cerebral palsy. The scale involves passively moving a limb through its range of motion and evaluating the resistance felt. The scoring ranges from 0 to 4, where 0 indicates no increase in muscle tone, 1 represents a slight increase with a catch or minimal resistance at the end of the range, and 1+ reflects a catch followed by minimal resistance through less than half of the movement. A score of 2 denotes a more marked increase in tone through most of the range, but the limb remains movable. 3 indicates considerable resistance, making movement difficult, and 4 signifies a rigid limb with severe spasticity. This scale is widely used in rehabilitation to monitor spasticity and guide treatment interventions.
Brunnstrom | Assessments will be conducted immediately before the treatment starts and at the end of the treatment (week 4).
  The Brunnstrom Stages of Recovery describe the six stages of motor recovery following a stroke or brain injury. In Stage 1, there is flaccidity, with no voluntary movement or reflex activity in the affected limb. Stage 2 marks the beginning of spasticity, with the emergence of basic limb synergies and minimal voluntary movement. In Stage 3, spasticity reaches its peak, and voluntary control is limited to synergy patterns. Stage 4 involves a decrease in spasticity, with the appearance of some voluntary movements outside of synergy patterns. By Stage 5, spasticity continues to decline, and more complex and isolated movements become possible. Finally, in Stage 6, normal movement patterns are largely restored, with minimal or no spasticity and full control of isolated joint movements.

CONTACTS AND LOCATIONS:
Overall Officials: Eda Gürçay, Prof., Study Director — Gaziler Physical Medicine and Rehabilitation Education and Research Hospital
Locations (1):
- SBÜ Gaziler Fizik Tedavi ve Rehabilitasyon Eğitim ve Araştırma Hastanesi, Ankara, Ankara, Turkey (Türkiye)